CLINICAL TRIAL: NCT03085134
Title: Clinical Safety & Efficacy of a New Infant Formula With Specific Medical Purpose (FSMP) Containing 2 Human Milk Oligosaccharides (HMOs)
Brief Title: Clinical Safety & Efficacy of a New Infant Formula With Specific Medical Purpose Containing Human Milk Oligosaccharides
Acronym: CINNAMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16.08.CLI
Record Dates: First submitted 2017-02-28; First posted 2017-03-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Health Maintenance Organizations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test infant formula with HMOs (Experimental): Extensively hydrolysed infant formula with HMOs taken by infant according to age, weight and appetite.
  Interventions: Other: Test infant formula with HMOs
- Control infant formula without HMOs (Active Comparator): Extensively hydrolysed infant formula without HMOs taken by infant according to age, weight and appetite
  Interventions: Other: Control infant formula without HMOs

INTERVENTIONS:
Other: Test infant formula with HMOs — Extensively hydrolysed (whey protein) specialty infant formulas (FSMP) with HMOs intended for management of CMPA.
  Arms: Test infant formula with HMOs
Other: Control infant formula without HMOs — Extensively hydrolysed (whey protein) specialty infant formulas (FSMP) intended for management of CMPA.
  Arms: Control infant formula without HMOs

SUMMARY:
The primary objective of the study is to show that infants with cow milk protein allergy (CMPA) fed with a new FSMP infant formula with reduced level of protein & with 2 Human Milk Oligosaccharides (HMOs) (test formula) have a growth in line with infants fed with a comparable FSMP formula but without HMOs (control formula). The secondary objectives are to assess whether consumption of Test formula by CMPA infants (i) reduces medication use and risk for infections in particular lower respiratory tract infections/morbidity, (ii) is well tolerated and allows for age appropriate growth and (iii) reduces health care costs.

DETAILED DESCRIPTION:
Infants with physician diagnosed CMPA, aged between birth and 6 months of age will take either the control or new test infant formula for 4 months and if judged suitable by physician, up to maximum of 12 months of age. Growth, adverse events, medication use and tolerance to formula will be assessed. As part of exploratory objectives, the study will also explore possible mode of action of the Test formula in CMPA infants, by assessing whether consumption of Test formula by CMPA infants affects stool microbiota and metabolic signatures as well as urine metabolic signatures and whether such changes can be associated to the intestinal inflammatory/health status, and the clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. Full term infant (37 weeks ≤ gestation ≤ 42 weeks)
2. 2500g ≤ birth weight ≤ 4500g
3. Written informed consent.
4. Infant aged between birth and 6 months.
5. Not being breastfed at time of enrollment or mothers of CMPA infant doing breastfeeding and independently elected before enrollment to exclusively formula feed.
6. Infants with physician diagnosed (and untreated with extensively hydrolysed or amino acid infant formula) Cow Milk Protein Allergy as per standard clinical practice and with at least 2 protocol specified symptoms present.

Exclusion Criteria:

1. Prior treatment with extensively hydrolysed infant formula for more than 72 hours or with amino acid infant formula.
2. Congenital illness or malformation that may affect growth.
3. Demonstrated chronic malabsorption not due to CMPA.
4. Significant pre-natal and/or serious post-natal disease other than CMPA before enrollment (per investigator's medical decision).
5. Minor parent(s).
6. Infants whose parents or caregivers cannot be expected to comply with study procedures.
7. Currently participating or having participated in another clinical trial since birth.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Growth expressed as weight gain in grams per day | 4 months
  Body weight measured from enrollment to 4 months of study formula intake

SECONDARY OUTCOMES:
Safety and medication use | 12 months
  Assessment of occurrence of adverse events (Number of adverse events per infant and number of infants with adverse events) and use of concomitant medication (specifically amount of antipyretics and antibiotics used per infant and number of infants using these) from enrollment until infants are 12 months of age.
Growth in terms of body weight. | 12 months
  Body weight (in kilograms) measured from enrollment until infants are 12 months of age.
Growth in terms of body length | 12 months
  Body length (in centimetres) measured from enrollment until infants are 12 months of age.
Growth in terms of head circumference | 12 months
  Head circumference (in centimetres) measured from enrollment until infants are 12 months of age.
Digestive tolerance and alleviation of CMPA | 12 months
  Recording of stool characteristics and frequency in diary, assessment of infant behavior pattern and medical assessment at each visit from enrollment until last study formula intake. Outcome will be reported as score on CoMiSS tool.
Compliance to study formula intake | 12 months
  Recording daily quantity consumed (in milliliters) in feeding diary for 3 days immediately before each visit from enrollment until last study formula intake.
Healthcare resource use assessed with Questionnaire | 12 months
  Questionnaire completed from enrollment until infants are 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Olesen, Study Chair — Nestlé Health Science Spain
Locations (42):
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - University Hospital Brussels, Brussels
  - CHC clinique de l'Esperance, Montegnée
- Hungary (3):
  - Clinexpert Gyogycentrum, Budapest
  - Bagoly Egeszseghaz, Kecskemét
  - Csolnoky Ferenc Korhaz, Veszprém
- Italy (5):
  - A.O.U Ospedali Riuniti, Ancona
  - Ospedale Luigi Sacco, Polo Universitario, Milan
  - University of Naples Federico II, Naples
  - A.O.U.P - Università degli Studi di Palermo, Palermo
  - University of Rome La Sapienza, Roma
- Poland (9):
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny Anna Ploszczuk, Bialystok
  - Specjalistyczna Przychodnia Lekarska Medicus, Chorzów
  - Gdańskie Centrum Zdrowia Sp. z o.o., Gdansk
  - NZOZ Medicus, Gostynin
  - ATOPIA - Specjalistyczna Przychodnia Medyczna, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Alergo-Med Specjalistyczna Przychodnia Lekarska SP. Z.O.O, Tarnów
  - Centrum Medyczne Lucyna Andrzej Dymek NZOZ S.C., Zawadzkie
- Singapore (4):
  - KK Women's and Children's Hospital, Singapore
  - Mount Elizabeth Medical Centre - Chiang Children's Allergy & Asthma Clinic, Singapore
  - Mount Elizabeth Medical Centre - The Child and Allergy Clinic, Singapore
  - National University Hospital, Singapore
- Spain (6):
  - Hospital Teresa Herrera, A Coruña
  - Hospital de Poniente, Almería
  - EBA Centelles, Barcelona
  - Hospital de Nens, Barcelona
  - Hospital Quirónsalud, Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
- United Kingdom (12):
  - Buckinghamshire Healthcare NHS Trust, Stoke Mandeville Hospital, Aylesbury
  - Northern Devon Healthcare NHS Trust, North Devon District Hospital, Barnstaple
  - Burton Hospitals NHS Foundation Trust, Queen's Hospital, Burton-on-Trent
  - Epsom and St Helier University Hospitals NHS Trust, St Helier University Hospital, Carshalton
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Medway NHS Foundation Trust, Medway Maritime Hospital, Gillingham
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Queen Elizabeth Hospital, King's Lynn NHS Foundation Trust, Kings Lynn
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No